CLINICAL TRIAL: NCT07042542
Title: The Effect of the Mulligan Spinal Mobilization Technique With Arm Movement on Pain, Grip Strength, and Functionality in Individuals With Carpal Tunnel Syndrome
Brief Title: Mulligan Mobilization With Arm Movement in CTS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beste Gebologlu (Other)
Responsible Party: Sponsor-Investigator, Beste Gebologlu, Physiotherapist and Graduate Student Researcher, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTS-MED25-BG; E-10840098-772.02-3960 (Other: Istanbul Medipol University Non-Interventional Clinical Research Ethics Committee)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Mulligan Spinal Mobilization with Arm Movement; Conventional Neurodynamic Mobilization; Functionality; Grip Strength; Rehabilitation; Pain; Median Nerve
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled parallel design comparing Mulligan mobilization with neurodynamic mobilization in patients with carpal tunnel syndrome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mulligan Spinal Mobilization with Arm Movement (Experimental): Participants in this group received Mulligan spinal mobilization applied to the cervical spine at C5, C6, and C7 levels, in 3 sets of 3 repetitions per level. During mobilization, participants actively performed arm movements in a neurodynamic stretching position. The intervention was administered 3 sessions per week for 6 weeks. Additionally, all participants performed tendon gliding and hand strengthening exercises three times per week for 6 weeks, which were also prescribed as home-based programs.
  Interventions: Other: Mulligan Spinal Mobilization with Arm Movement; Behavioral: Tendon Gliding and Hand Strengthening Exercises
- Conventional Neurodynamic Mobilization (Active Comparator): Participants in this group received conventional neurodynamic mobilization techniques targeting the median nerve, applied by a therapist. The intervention was administered 3 sessions per week for 6 weeks, with 3 sets of 3 repetitions in each session. In addition, all participants performed tendon gliding exercises and hand strengthening exercises three times per week for 6 weeks. These exercises were also assigned as home-based programs.
  Interventions: Other: Conventional Neurodynamic Mobilization; Behavioral: Tendon Gliding and Hand Strengthening Exercises

INTERVENTIONS:
Other: Mulligan Spinal Mobilization with Arm Movement — In the neurodynamic SNAGs technique, participants sat on a chair. The therapist placed the medial border of the distal phalanx of one thumb under the facet joints of the C5, C6, and C7 levels, respectively. Then, the therapist placed the tip of the other thumb on the lateral side of the first thumb. In neurodynamic spinal mobilization combined with arm movement, the therapist provided manual contact to the affected spinous process level by supporting the medial aspect of one thumb with the index finger of the other hand. The therapist applied a transverse shift from the affected side to the unaffected side, but only in the transverse plane. While the glide was in progress, the patient was asked to perform neurodynamic movements for the median nerve, including scapular depression, shoulder abduction, elbow extension, forearm supination, and wrist and finger extension, all without crossing the pain limit for the affected side.
  Arms: Mulligan Spinal Mobilization with Arm Movement
Other: Conventional Neurodynamic Mobilization — A neurodynamic mobilization technique involving a specific sequence of movements along the median nerve line was applied. For the right side, the procedure was performed as follows: The individual was placed supine on a stretcher. The therapist stood on the right side of the stretcher, facing the participant, with their right leg in front of their left leg. The individual's arm rested on the therapist's right thigh, and the therapist held the individual's right hand with his left hand. During the procedure, the therapist placed one hand on the individual's shoulder to depress the shoulder girdle by pressing the scapula downward. The individual's shoulder was abducted 90° and laterally rotated, and the forearm was supinated. The wrist, thumb, and fingers were extended. In this position, the therapist dynamically alternated between simultaneous elbow flexion/wrist extension and simultaneous elbow extension/wrist flexion.
  Arms: Conventional Neurodynamic Mobilization
Behavioral: Tendon Gliding and Hand Strengthening Exercises — Tendon glide exercises were performed in five consecutive positions. Each position was practiced for seven seconds, with three sets of five repetitions and one minute of rest between sets. Participants were asked to perform the exercises three times during the day. Hand muscle strengthening exercises were performed by placing a tire on the fingertips, abducting the fingers, and stretching the tire to strengthen the intrinsic muscles and fingers. Resistance could be increased by thickening the tire or adding a second one. Participants were given a grip strength exercise. The hand grip exercise strengthened the extrinsic muscles. Finger flexion and extension exercises strengthened the hand and finger muscles. Participants were asked to perform 10 repetitions of each exercise in each session and to perform the strengthening exercises three times during the day.

SUMMARY:
The aim of this study was to investigate the effect of the Mulligan Spinal Mobilization with Arm Movement technique on pain, grip strength and functionality in individuals with carpal tunnel syndrome and to compare it with the conventional neurodynamic mobilization technique. The study aims to answer the following questions:

Is the Mulligan spinal mobilization technique with arm movement superior to the conventional neurodynamic mobilization technique in terms of pain, grip strength, and functionality in individuals with carpal tunnel syndrome? Does the Mulligan spinal mobilization technique with arm movement outperform the conventional neurodynamic mobilization technique in terms of pain, grip strength, and functionality in individuals with carpal tunnel syndrome? The evaluation process took place in three stages for both groups: Baseline (pre-test), 6 weeks after the start of the study (post-test), and 12 weeks after the start of the study (follow-up test).

DETAILED DESCRIPTION:
Thirty participants completed the randomized controlled trial and were divided into two groups as the study group (Mulligan group) and the control group (conventional neurodynamic mobilization). Both groups received tendon gliding exercises (TGE) and strengthening exercises for the intrinsic and extrinsic muscles of the hand during the treatment period. The treatment period lasted six weeks, and after the end of the treatment, the individuals were followed up with a home program until the 12th week. Evaluations were performed three times at baseline, 6 and 12 weeks and included measures of pain (VAS, McGill), functionality (DASH, FDS, FDS), grip strength (Jamar hand dynamometer), range of motion and sensation (Semmes-Weinstein monofilament test). The control group received Mulligan's neurodynamic spinal mobilisation technique at the C5-C6-C7 levels with arm movement for six weeks. This involved three sessions per week, each comprising three sets of three repetitions, with each repetition lasting an average of one minute. The total duration of each session was approximately ten minutes.

The control group received the same technique without the Mulligan approach for six weeks, three days a week, three sets of three repetitions, with each repetition lasting an average of one minute. After the treatment period, both groups performed a standard exercise programme consisting of tendon gliding and hand strengthening exercises, which were also recommended to patients at the end of each session. These exercises were continued throughout the follow-up period after treatment.

The study was completed between June 2023 and January 2025 with ethical approval from Istanbul Medipol University.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of mild to moderate carpal tunnel syndrome (CTS).
* Being between 20 and 60 years of age.
* Having symptoms of paresthesia, pain, and numbness in areas of the hand related to the median nerve lasting more than six weeks.
* A positive Tinel, Phalen, or carpal compression test during wrist examination.

Exclusion Criteria:

* Pregnancy.
* The patient has a contraindication to exercise.
* Additional neurological, rheumatological, and orthopedic conditions.
* A positive Spurling test.
* Patients who have undergone surgery in the wrist or neck region.
* Presence of a tumor or pathology in the cervical region.
* Patients who have received physical therapy for the wrist or neck in the last six months.
* The patient has mental health issues.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline, 6th week, 12th week
  Pain intensity was assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst pain), at rest and during activity with higher scores indicating worse pain.
Functional Status and Symptom Severity | Baseline, 6th week, 12th week
  Functional status and symptom severity were evaluated using the Boston Carpal Tunnel Questionnaire, including the Functional Status Scale (FSS) and Symptom Severity Scale (SSS). Each scale ranges from 1 to 5. Higher scores indicate greater disability (FSS) or more severe symptoms (SSS).

SECONDARY OUTCOMES:
Hand Grip Strength | Baseline, 6th week, 12th week
  Hand grip strength was measured using a dynamometer in kilograms to assess functional improvement. There is no fixed scoring range; higher values indicate greater muscle strength and improved function.
Range of Motion of the Wrist | Baseline, 6th week, 12th week
  Wrist range of motion was measured in degrees using a goniometer, including supination, pronation, radial deviation, ulnar deviation, flexion, and extension. There is no fixed scale; higher degrees represent greater joint mobility.
Sensory Function | Baseline, 6th week, 12th week
  Sensory function was evaluated using the Semmes-Weinstein monofilament test on the median nerve-innervated area. Filaments of varying thickness were used to determine sensory threshold. Lower values indicate greater sensitivity, while higher filament values indicate decreased sensory function.
Pain Quality - McGill Pain Questionnaire | Baseline, 6th week, 12th week
  Pain quality and intensity were assessed. The McGill Pain Questionnaire scores range from 0 to 78. Higher scores indicate worse pain experience.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar KAYA SARIBAS, Assoc Prof, Principal Investigator — Istanbul Medipol University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Istanbul Medipol University, Istanbul, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a non-commercial academic thesis study and there is no plan to share individual participant data (IPD) with other researchers.